CLINICAL TRIAL: NCT05892666
Title: The Right Care, for the Right Patient, at the Right Time, by the Right Provider: A Value-based Comparison of the Management of Ambulatory Patients With Acute Health Concerns in walk-in Clinics, Primary Care Physician Practices and Emergency Departments
Status: Recruiting | Type: Observational
Sponsor: Simon Berthelot (Other)
Responsible Party: Sponsor-Investigator, Simon Berthelot, Emergency Physician, CHU de Québec-Université Laval; Associate Professor, Faculté of medicine, Université Laval, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Other Study IDs: Value trial
Record Dates: First submitted 2023-05-01; First posted 2023-06-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Ambulatory Care; Emergency Services, Hospital; Quality of Care; Costs
MeSH Terms: conditions — Emergencies | interventions — Consent Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Emergency department: ED care for acute ambulatory conditions by physicians unfamiliar with the patients.
  Interventions: Other: On-site recruitment (information and consent) following a random sampling recruitment schedule; Other: First phone call 1-3 days after the initial visit; Other: Second phone call 8-14 days after the initial visit
- Walk-in clinics: In-person or virtual care in a walk-in clinic for acute ambulatory conditions by physicians unfamiliar with the patients. In-person and virtual care will be assessed together as part of the care offer in outpatient clinics, but separately as a sub-analysis.
  Interventions: Other: On-site recruitment (information and consent) following a random sampling recruitment schedule; Other: First phone call 1-3 days after the initial visit; Other: Second phone call 8-14 days after the initial visit
- Primary care practice: In-person or virtual care in a primary care clinic for acute ambulatory conditions (patients attached to a primary care practice, seen by their family physician or a colleague on a same-day appointment for urgent needs). In-person and virtual care will be assessed together as part of the care offer in outpatient clinics, but separately as a sub-analysis.
  Interventions: Other: On-site recruitment (information and consent) following a random sampling recruitment schedule; Other: First phone call 1-3 days after the initial visit; Other: Second phone call 8-14 days after the initial visit

INTERVENTIONS:
Other: On-site recruitment (information and consent) following a random sampling recruitment schedule — A trained research assistant in collaboration with local clerks at each site will screen eligible patients after on-site registration or online scheduling, but prior to assessment by a physician, based on included presenting complaints. The research assistant or member of the care team, depending on the local rules, will approach the potentially eligible participants and present them the research project and information consent form. If the patient agrees to participate and is eligible, they will sign the information and consent form and the research assistant will take their vital signs (for onsite participants only).
Other: First phone call 1-3 days after the initial visit — Once the patient has been discharged, a research assistant will call the patient within 72 hours following the initial visit. This phone call will allow to i) ensure that gender, ethnicity, comorbidities and disposition plans are fully documented; and ii) use our patient-reported experience measure tool and administer a questionnaire on motivation for choosing one care setting over the other. Motivation will be classified in the 6 domains of the Conceptual Model of Emergency Department Use (Uscher-Pines et al. 2019). Participants will be asked to specify whether their choice of care setting was based on accessibility, convenience, their perception of the severity of illness, their beliefs and knowledge regarding these care settings, referral/advice from a care professional or an acquaintance, or on costs.
Other: Second phone call 8-14 days after the initial visit — A follow-up phone call will be made to all participants 8 days after the initial visit to evaluate primary and secondary outcome metrics. Patient-reported outcome (primary) and cost measures will be completed by the participants at this moment.

SUMMARY:
INTRODUCTION Whereas low-acuity ambulatory patients have been cited as a source of emergency department (ED) overuse or misuse, it is argued that patient evaluation in the ED may end up being more cost-effective. The COVID-19 pandemic has complicated the debate by shifting primary care practices (PCP) and walk-in clinics (WIC) towards telemedicine, a consultation modality presumed to be more efficient under the circumstances.

OBJECTIVES To compare, from patient and healthcare system perspectives, the value of the care received in person or by telemedicine in EDs, WICs and PCPs by ambulatory patients presenting with one the following complaints: 1) Acute diarrheas; 2) Sore throat; 3) Nasal congestion; 4) Increased or purulent nasal discharge; 5) Earache or ear discharge; 6) Shortness of breath; 7) Cough; 8) Increased or purulent sputum; 9) Muscle aches; 10) Anosmia; 11) Dysgeusia; 12) Burning urine; 13) Urinary frequency and urgency; 14) Dysuria; 15) Limb traumatic injury; 16) Cervical, thoracic or lumbar back pain; and 17) Fever

METHODS The investigators shall perform a multicenter prospective cohort study in Québec and Ontario. In phase 1, a time-driven activity-based costing method will be applied at each of 14 study sites. This method uses time as a cost driver to allocate direct costs (e.g. medication), consumable expenditures (e.g. needles, office supplies), overhead (e.g. building maintenance) and physician charges to patient care. The cost of a care episode thus will be proportional to the time spent receiving the care. At the end of this phase, a list of care process costs (e.g. triage, virtual medical assessment) will be generated and used to calculate the cost of each consultation during phase 2, in which a prospective cohort of patients will be monitored in order to compare the care received in EDs, WICs and PCPs. Research assistants will recruit eligible participants during the initial in-person or virtual visit. They will complete the collection using local medical records and provincial databases. Participants will be contacted by phone for follow-up questionnaires 1-3 and 8-14 days after their visit. Patients shall be aged 18 years and over, ambulatory throughout the care episode and have one of the targeted presenting complaints mentioned above. The estimated sample size is 3,906 patients. The primary outcome measurement for comparing the three types of care setting will be patient-reported outcome scores. The secondary outcome measurements will be: 1) patient-reported experience scores; 2) mean costs borne wholly by patients; 3) the proportion of return visits to any site 3 and 7 days after the initial visit; 4) the mean cost of care; 5) the incidences of mortality, hospital admissions and placement in intensive care within 30 days following the initial visit; 6) adherence to practice guidelines. Multilevel generalized linear models will be used to compare the care setting types and an overlap weights approach will be applied to adjust for confounding due to age, sex, gender, ethnicity, comorbidities, registration with a family physician, socioeconomic status and perceived severity of illness.

EXPERTISE This research project brings together a strong team with expertise in emergency and primary care, pneumonology, performance assessment, biostatistics, health economics, patient-oriented research, knowledge translation, administration and policymaking.

IMPORTANCE The endpoint of our program will be for policymakers, patients and care providers to be able to determine the most appropriate care setting for the management of ambulatory emergency conditions, based on the value of care associated with each alternative.

ELIGIBILITY:
We shall include patients:

1. aged 18 years and over;
2. seen in person or via telemedicine in an ED, a walk-in clinic, or the primary care practice where they are registered;
3. ambulatory during the entire visit or consultation;
4. with one of the following presenting complaints:

   1. acute diarrheas, defined as at least one day (24h) reported with three or more loose or liquid stools in the last seven days;
   2. Sore throat;
   3. Nasal congestion;
   4. Increased or purulent nasal discharge;
   5. Earache or ear discharge;
   6. Shortness of breath;
   7. Cough;
   8. Increased or purulent sputum;
   9. Muscle aches;
   10. Anosmia;
   11. Dysgeusia;
   12. Burning urine;
   13. Urinary frequency and urgency;
   14. Dysuria;
   15. Limb traumatic injury;
   16. Cervical, thoracic or lumbar back pain;
   17. Fever.

We shall exclude patients:

1. transported by ambulance;
2. not covered by the provincial health insurance plan;
3. having consulted for a similar problem in the previous 30 days since patients with refractory disease represent a population with different care needs.;
4. living in a long-term healthcare facility or incarcerated;
5. with cognitive impairment that prevents reliable answers to the research questions;
6. receiving palliative care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our assessment will focus on patients presenting with acute ambulatory conditions, which share the common feature of being potentially treatable in EDs, walk-in clinics or primary care practices.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Median PROM-ED scores | At 7 days after the initial visit measured at the 8-14 day follow-up call
  The adapted PROM-ED provides a measurement of patient-reported outcome expressed as scores for symptom relief, reassurance and having a plan for care. Responses for each dimension are aggregated reported as a percentage, with a higher percentage signifying better health outcomes according to the patient

SECONDARY OUTCOMES:
Patient-reported experience measure (PREM) scores | At the end of the initial visit measured at the 1-3 day follow-up call
  The PREM evaluates the patient's view of care delivery and measures various dimensions of patient experience (e.g., attitude of providers). The main question for this primary outcome measure will be: "Would you recommend this place to your friends and family"? Most PREM questions are on a 5-level Likert scale.
Mean cost of disease for patients (CoPaQ) | At 7 days measured at the 8-14 day follow-up call
  The adapted CoPaQ measures patients' and caregivers' out-of-pocket expenses (e.g., travel) and indirect costs (e.g., loss of income).
Incidence of return visit | At 7 days after the initial visit
  Proportion of patients returning to any ED or outpatient clinic at 72 h and 7 days after the initial visit. Return visit occurrences will be identified via provincial physician billing databases.
Mean cost of care - Health care system perspective | At 72 hours and 7 days after the initial visit
  Cost per care episode from the public payer's perspective calculated by summing the costs of all care processes delivered to a patient during the initial visit plus the costs of return visits and/or admissions at 72 hours and 7 days. Costs will be measured with a time-driven activity-based costing method with data extracted from electronic medical records review and provincial billing databases.
Incidences of admission/intensive care unit/mortality | At 7 and 30 days after the initial visit
  Proportions of patients who were admitted to hospital or to the intensive care unit or died within 30 days after the initial visit. Obtained via electronic medical records review and provincial databases (Institut de la statistique du Québec and ICES).
Wait times | For the initial visit
  Median/mean length of stay and time spent waiting to see a physician obtained via electronic medical records
Incidence of oral corticosteroid prescription | For the initial visit
  Proportion of patients with exacerbated asthma or COPD who received a prescription for oral corticosteroids. Obtained via electronic medical records
Incidence of antibiotic or antiviral medication prescription | For the initial visit
  Proportions of patients with URTI, otitis media, influenza or bronchitis who received a prescription for antibiotics or antiviral medication. Obtained via electronic medical records.
Incidence of narcotic prescription | For the initial visit
  Proportions of patients with cervical, thoracic and lumbar back pain who received a prescription for narcotics. Obtained via electronic medical records.
Incidence of chest X-ray use | For the initial visit
  Proportions of patients with URTI, bronchitis, asthma and back pain who had a chest X-ray performed. Obtained via electronic medical records.
Incidence of spine X-ray, CT scan or MRI use | For the initial visit
  Proportions of patients with back pain who had a spine X-ray, CT scan or a magnetic resonance imaging (MRI) performed or prescribed. Obtained via electronic medical records.
Compliance to guidelines on use of antibiotics | For the initial visit
  Proportions of compliance to provincial recommendations of antibiotic prescriptions for pneumonia, tonsillitis, acute exacerbation of COPD and urinary tract infection. Obtained via electronic medical records.
Incidence of diagnostic spirometry prescription | For the initial visit
  Proportions of spirometry prescribed for long-term >40-year-old smokers (current or past) undiagnosed with COPD who present for an acute lower respiratory tract infection. Obtained via electronic medical records.
Mean greenhouse gas (GHG) emissions from patient transportation to consultation site | For the initial visit
  Calculated following the Québec Ministry of Environment "Guide to quantifying greenhouse gas emissions". Fuel consumption (in liters) will be estimated from patient transport modality and travel distance (in km) between home and consultation site. GHS emissions in kg of CO2 equivalent will be calculated by multiplying fuel consumption (L) by the appropriate emission coefficient (kg CO2 eq./L) depending on the transport modality used (e.g. car, bus). Distance obtained at the 8-14 day follow-up call.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Berthelot, MD MSc FRCPC CCMF(MU), Principal Investigator — CHU de Québec-Université Laval; Mylaine Breton, PhD, Principal Investigator — Université de Sherbrooke; Jason R. Guertin, PhD, Principal Investigator — Laval University
Locations (7):
- Canada (7):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Queen's Family Health Team, Kingston, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - CISSS de Lanaudière, Joliette, Quebec
  - CIUSSS-Nord de Montréal, Montreal, Quebec
  - CIUSSS de la Capitale-Nationale, Québec
  - Centre de recherche CHU de Québec - Université Laval, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berthelot S, Breton M, Guertin JR, Archambault PM, Berger Pelletier E, Blouin D, Borgundvaag B, Duhoux A, Harvey Labbe L, Laberge M, Lachapelle P, Lapointe-Shaw L, Layani G, Lefebvre G, Mallet M, Matthews D, McBrien K, McLeod S, Mercier E, Messier A, Moore L, Morris J, Morris K, Ovens H, Pageau P, Paquette JS, Perry J, Schull M, Simon M, Simonyan D, Stelfox HT, Talbot D, Vaillancourt S. A Value-Based Comparison of the Management of Ambulatory Respiratory Diseases in Walk-in Clinics, Primary Care Practices, and Emergency Departments: Protocol for a Multicenter Prospective Cohort Study. JMIR Res Protoc. 2021 Feb 22;10(2):e25619. doi: 10.2196/25619. PMID 33616548